CLINICAL TRIAL: NCT00069472
Title: Genetics of Rheumatoid Arthritis Registry
Brief Title: Genetic Registry for Rheumatoid Arthritis
Acronym: NARAC
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Arthritis Foundation (Other)
Responsible Party: Principal Investigator, Peter Gregersen, Center Head, Robert S Boas Center for Genomics and Human Genetics, Northwell Health
Other Study IDs: NIAMS-107; N01AR72232-001 (NIH)
Record Dates: First submitted 2003-09-25; First posted 2003-09-29 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Genetics
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA, plasma, serum and cells
Oversight: Data Monitoring Committee: No

SUMMARY:
Many genes are thought to contribute to rheumatoid arthritis (RA). This study will attempt to identify genes that may contribute to RA.

DETAILED DESCRIPTION:
The identification of genes for complex disorders such as RA requires large numbers of genetically informative families. This study enrolls people diagnosed with with RA and their families.

This study will enroll 1000 RA patients and their parents. Participants with RA will be evaluated at his or her doctor's office or other location convenient for the participant. Participants will have a brief phone interview with a study coordinator and a blood sample will be obtained. Disease evaluation will be done at one visit and will include confirmation of diagnosis, a 28 joint count, joint alignment and mobility score (JAMS) and administration of a health assessment questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adult onset RA
* Diagnosis of RA made between 18 and 60 years old
* Both parents alive and willing to participate
* Parents may have diagnosis of RA (affected) or be unaffected

Exclusion Criteria:

* Inflammatory bowel disease
* Lupus
* Psoriatic arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with RA who have two living biological parents. Parents can be affected or unaffected with RA. We call the family units "trios".
Sampling Method: Non-Probability Sample
Enrollment: 1062 (Actual)
Dates: Start 2002-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Genetic Association with risk for rheumatoid arthritis | 10 years
  The project aims to identify risk alleles for rheumatoid arthritis using association methods in trio families, combined with data from singleton cases and multiplex families

CONTACTS AND LOCATIONS:
Overall Officials: Peter K. Gregersen, MD, Principal Investigator — North Shore University Hospital
Locations (1):
- Feinstein Institute for Medical Research, Manhasset, New York, United States

REFERENCES:
- [Background] Jawaheer D, Li W, Graham RR, Chen W, Damle A, Xiao X, Monteiro J, Khalili H, Lee A, Lundsten R, Begovich A, Bugawan T, Erlich H, Elder JT, Criswell LA, Seldin MF, Amos CI, Behrens TW, Gregersen PK. Dissecting the genetic complexity of the association between human leukocyte antigens and rheumatoid arthritis. Am J Hum Genet. 2002 Sep;71(3):585-94. doi: 10.1086/342407. Epub 2002 Aug 9. PMID 12181776
- [Background] Jawaheer D, Seldin MF, Amos CI, Chen WV, Shigeta R, Monteiro J, Kern M, Criswell LA, Albani S, Nelson JL, Clegg DO, Pope R, Schroeder HW Jr, Bridges SL Jr, Pisetsky DS, Ward R, Kastner DL, Wilder RL, Pincus T, Callahan LF, Flemming D, Wener MH, Gregersen PK. A genomewide screen in multiplex rheumatoid arthritis families suggests genetic overlap with other autoimmune diseases. Am J Hum Genet. 2001 Apr;68(4):927-36. doi: 10.1086/319518. Epub 2001 Mar 9. PMID 11254450
- [Background] Jawaheer D, Seldin MF, Amos CI, Chen WV, Shigeta R, Etzel C, Damle A, Xiao X, Chen D, Lum RF, Monteiro J, Kern M, Criswell LA, Albani S, Nelson JL, Clegg DO, Pope R, Schroeder HW Jr, Bridges SL Jr, Pisetsky DS, Ward R, Kastner DL, Wilder RL, Pincus T, Callahan LF, Flemming D, Wener MH, Gregersen PK; North American Rheumatoid Arthritis Consortium. Screening the genome for rheumatoid arthritis susceptibility genes: a replication study and combined analysis of 512 multicase families. Arthritis Rheum. 2003 Apr;48(4):906-16. doi: 10.1002/art.10989. PMID 12687532
- [Background] Eyre S, Bowes J, Diogo D, Lee A, Barton A, Martin P, Zhernakova A, Stahl E, Viatte S, McAllister K, Amos CI, Padyukov L, Toes RE, Huizinga TW, Wijmenga C, Trynka G, Franke L, Westra HJ, Alfredsson L, Hu X, Sandor C, de Bakker PI, Davila S, Khor CC, Heng KK, Andrews R, Edkins S, Hunt SE, Langford C, Symmons D; Biologics in Rheumatoid Arthritis Genetics and Genomics Study Syndicate; Wellcome Trust Case Control Consortium; Concannon P, Onengut-Gumuscu S, Rich SS, Deloukas P, Gonzalez-Gay MA, Rodriguez-Rodriguez L, Arlsetig L, Martin J, Rantapaa-Dahlqvist S, Plenge RM, Raychaudhuri S, Klareskog L, Gregersen PK, Worthington J. High-density genetic mapping identifies new susceptibility loci for rheumatoid arthritis. Nat Genet. 2012 Dec;44(12):1336-40. doi: 10.1038/ng.2462. Epub 2012 Nov 11. PMID 23143596
- [Background] Raychaudhuri S, Sandor C, Stahl EA, Freudenberg J, Lee HS, Jia X, Alfredsson L, Padyukov L, Klareskog L, Worthington J, Siminovitch KA, Bae SC, Plenge RM, Gregersen PK, de Bakker PI. Five amino acids in three HLA proteins explain most of the association between MHC and seropositive rheumatoid arthritis. Nat Genet. 2012 Jan 29;44(3):291-6. doi: 10.1038/ng.1076. PMID 22286218
- [Background] Gregersen PK, Amos CI, Lee AT, Lu Y, Remmers EF, Kastner DL, Seldin MF, Criswell LA, Plenge RM, Holers VM, Mikuls TR, Sokka T, Moreland LW, Bridges SL Jr, Xie G, Begovich AB, Siminovitch KA. REL, encoding a member of the NF-kappaB family of transcription factors, is a newly defined risk locus for rheumatoid arthritis. Nat Genet. 2009 Jul;41(7):820-3. doi: 10.1038/ng.395. Epub 2009 Jun 7. PMID 19503088
- [Background] Plenge RM, Seielstad M, Padyukov L, Lee AT, Remmers EF, Ding B, Liew A, Khalili H, Chandrasekaran A, Davies LR, Li W, Tan AK, Bonnard C, Ong RT, Thalamuthu A, Pettersson S, Liu C, Tian C, Chen WV, Carulli JP, Beckman EM, Altshuler D, Alfredsson L, Criswell LA, Amos CI, Seldin MF, Kastner DL, Klareskog L, Gregersen PK. TRAF1-C5 as a risk locus for rheumatoid arthritis--a genomewide study. N Engl J Med. 2007 Sep 20;357(12):1199-209. doi: 10.1056/NEJMoa073491. Epub 2007 Sep 5. PMID 17804836
- [Background] Remmers EF, Plenge RM, Lee AT, Graham RR, Hom G, Behrens TW, de Bakker PI, Le JM, Lee HS, Batliwalla F, Li W, Masters SL, Booty MG, Carulli JP, Padyukov L, Alfredsson L, Klareskog L, Chen WV, Amos CI, Criswell LA, Seldin MF, Kastner DL, Gregersen PK. STAT4 and the risk of rheumatoid arthritis and systemic lupus erythematosus. N Engl J Med. 2007 Sep 6;357(10):977-86. doi: 10.1056/NEJMoa073003. PMID 17804842